CLINICAL TRIAL: NCT00066703
Title: A Phase III Trial Evaluating The Role Of Exemestane Plus GnRH Analogue As Adjuvant Therapy For Premenopausal Women With Endocrine Responsive Breast Cancer
Brief Title: Triptorelin With Either Exemestane or Tamoxifen in Treating Premenopausal Women With Hormone-Responsive Breast Cancer
Acronym: TEXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Breast International Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCSG 25-02 / BIG 3-02; IBCSG 25-02; BIG 3-02 (Other: Breast International Group); NABCI IBCSG 25-02; EU-20347; 2004-000168-28 (EudraCT Number); CDR0000316458 (Registry Identifier: CT.gov)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen; Triptorelin Pamoate; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- T+OFS (Active Comparator): Ovarian function suppression (OFS) by triptorelin (GnRH analogue) 3.75mg by im injection q28 days for 5 years plus tamoxifen 20mg orally daily for 5 years. Tamoxifen (T) begins after the completion of adjuvant chemotherapy if given, or approximately 6-8 weeks after the initiation of triptorelin. Bilateral oophorectomy or ovarian irradiation was allowed after at least 6 months of triptorelin.
  Interventions: Drug: tamoxifen; Drug: triptorelin
- E+OFS (Experimental): Ovarian function suppression (OFS) by triptorelin (GnRH analogue) 3.75mg by im injection q28 days for 5 years plus exemestane 25mg orally daily for 5 years. Exemestane (E) begins after the completion of adjuvant chemotherapy if given, or approximately 6-8 weeks after the initiation of triptorelin. Bilateral oophorectomy or ovarian irradiation was allowed after at least 6 months of triptorelin.
  Interventions: Drug: exemestane; Drug: triptorelin

INTERVENTIONS:
Drug: exemestane
  Other Names: Aromasin
  Arms: E+OFS
Drug: tamoxifen
  Other Names: Nolvadex
  Arms: T+OFS
Drug: triptorelin
  Other Names: GnRH analogue; Trelstar Depot; Decapeptyl Depot

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using triptorelin, exemestane, and tamoxifen may fight breast cancer by blocking the use of estrogen. It is not yet known whether giving triptorelin together with exemestane is more effective than triptorelin and tamoxifen in treating hormone-responsive breast cancer.

PURPOSE: This randomized phase III trial is studying triptorelin and exemestane to see how well they work compared to triptorelin and tamoxifen in treating premenopausal women with hormone-responsive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival, breast cancer-free interval, distant recurrence-free interval and overall survival of premenopausal women with endocrine-responsive breast cancer when treated with triptorelin and exemestane vs triptorelin and tamoxifen.
* Compare the quality of life, including late side effects of early menopause, of patients treated with these regimens.

OUTLINE: This is a randomized, international, multicenter study. Patients are stratified according to planned use of concurrent adjuvant chemotherapy (yes vs no), and number of positive lymph nodes (0 vs 1 or more). Treatment duration is 5 years. Patients are followed every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter. Quality of life is assessed at baseline, every 6 months for 2 years, and annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer
* Completely resected disease

  * No clinically detectable residual loco-regional axillary disease
  * Prior surgery for primary breast cancer of 1 of the following types:

    * Total mastectomy with or without adjuvant radiotherapy
    * Breast-conserving procedure (e.g., lumpectomy, quadrantectomy, or partial mastectomy with margins negative* for invasive disease and ductal carcinoma in situ) with planned radiotherapy NOTE: *If all other margins are clear a positive posterior (deep) margin is permitted, provided the excision was performed down to the pectoral fascia and all tumor has been removed OR a positive anterior (superficial; abutting skin) margin is allowed provided all tumor was removed
* Tumor confined to the breast and axillary nodes

  * Tumor detected in internal mammary chain nodes by sentinel node procedure and is not enlarged is allowed
* Axillary lymph node dissection or a negative axillary sentinel node biopsy required

  * Patients with negative or microscopically positive axillary sentinel nodes are eligible
  * Positive sentinel nodes must have either axillary dissection or radiation of axillary nodes
* No distant metastases
* No locally advanced inoperable breast cancer, including any of the following:

  * Inflammatory breast cancer
  * Supraclavicular node involvement
  * Enlarged internal mammary nodes (unless pathologically negative)
* Bilateral synchronous invasive breast cancer allowed if disease meets all other eligibility criteria
* No prior ipsilateral or contralateral invasive breast cancer
* Hormone receptor status:

  * Estrogen and/or progesterone receptor positive

    * At least 10% of the tumor cells positive by immunohistochemistry
    * If > 1 breast tumor, each tumor must be hormone receptor positive

PATIENT CHARACTERISTICS:

Age

* Premenopausal

Sex

* Female

Menopausal status

* Premenopausal

  * Estradiol in the premenopausal range after prior surgery OR meets the following criteria:

    * Menstruating regularly for the past 6 months
    * Has not used any form of hormonal treatment (including hormonal contraception) within the past 6 months

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* No systemic hepatic disease that would preclude prolonged follow-up

Renal

* No systemic renal disease that would preclude prolonged follow-up

Cardiovascular

* No systemic cardiovascular disease that would preclude prolonged follow-up
* No prior thrombosis (e.g., deep vein thrombosis) and/or embolism unless patient is medically suitable

Pulmonary

* No systemic pulmonary disease that would preclude prolonged follow-up

Other

* Not pregnant or nursing
* Fertile patients must use effective nonhormonal contraception
* No history of noncompliance to medical regimens
* No other nonmalignant systemic disease that would preclude prolonged follow-up
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, nonbreast carcinoma in situ, contralateral or ipsilateral carcinoma in situ of the breast, or other nonrecurrent invasive nonbreast malignancy, including any of the following:

  * Stage I papillary thyroid cancer
  * Stage IA carcinoma of the cervix
  * Stage IA or B endometrioid endometrial cancer
  * Borderline or stage I ovarian cancer
* No psychiatric, addictive, or other disorder that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior or concurrent neoadjuvant or adjuvant trastuzumab allowed

Chemotherapy

* No prior neoadjuvant or adjuvant chemotherapy

Endocrine therapy

* No prior tamoxifen, other selective estrogen-receptor modulators (SERMs) (e.g., raloxifene), or hormone replacement therapy for more than 1 year before breast cancer diagnosis
* No prior neoadjuvant or adjuvant endocrine therapy since diagnosis of breast cancer
* No concurrent oral or transdermal hormonal therapy
* No other concurrent estrogen, progesterone, or androgens
* No other concurrent aromatase inhibitors
* No concurrent oral or other hormonal contraceptives (i.e., implants or depot injections)

Radiotherapy

* See Disease Characteristics
* No prior ovarian radiotherapy

Surgery

* See Disease Characteristics
* No prior bilateral oophorectomy

Other

* No concurrent bisphosphonates, except in the following cases:

  * Bone density is at least 1.5 standard deviations below the young adult normal mean
  * Participation in a randomized clinical study testing bisphosphonates in the adjuvant breast cancer setting
* No other concurrent investigational agents

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2672 (Actual)
Dates: Start 2003-11-03 (Actual); Primary Completion 2011-03-11 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Pagani, MD, Study Chair — Oncology Institute of Southern Switzerland; Barbara Walley, MD, FRCPC, Study Chair — Tom Baker Cancer Centre
Locations (228):
- United States (139):
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Ruby L. Golleher Cancer Program at Presbyterian Intercommunity Hospital, Whittier, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Kootenai Cancer Center - Coeur d'Alene, Coeur d'Alene, Idaho
  - Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Hospital, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Frederick Memorial Hospital Regional Cancer Therapy Center, Frederick, Maryland
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Bethke Cancer Center at Emerson Hospital, Concord, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Greenville, Greenville, South Carolina
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center at Erlanger Hospital - Baroness, Chattanooga, Tennessee
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Aurora Memorial Hospital of Burlington, Burlington, Wisconsin
  - Oncology Alliance - Franklin, Franklin, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Oncology Alliance - Kenosha South, Kenosha, Wisconsin
  - Aurora Advanced Healthcare East Mequon Clinic, Mequon, Wisconsin
  - Columbia-Saint Mary's Hospital-Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons Milwaukee, Mequon, Wisconsin
  - Oncology Alliance, SC - Milwaukee - South, Milwaukee, Wisconsin
  - Aurora Health Center - Racine, Racine, Wisconsin
  - Aurora Health Center - Waukesha, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
- Australia (20):
  - Cancer Therapy Centre at Campbelltown Hospital, Campbelltown, New South Wales
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Cancer Therapy Centre at Liverpool Hospital, Liverpool, New South Wales
  - Tamworth Base Hospital, Tamworth, New South Wales
  - Manning Base Hospital, Taree, New South Wales
  - Tweed Heads Hospital, Tweed Heads, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Breast Unit Mercy Private, East Melbourne, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St. Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Hutois, Huy
  - U.Z. Gasthuisberg, Leuven
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Centre Hospitalier Peltzer-La Tourelle, Verviers
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (9):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Trillium Health Centre - Mississauga Site, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Egypt (2):
  - Cairo Oncology Center, Cairo
  - National Cancer Institute of Egypt, Cairo
- Germany (15):
  - Brustzentrum Klinikum Mittelbaden, Baden-Baden
  - Klinikum Deggendorf, Deggendorf
  - Frauenklinik des Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsfrauenklinik Frankfurt, Frankfurt
  - Universitaets-Frauenklinik Goettingen, Göttingen
  - St. Vincentius - Kliniken, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Universitatsklinik Mainz, Mainz
  - Universitaetsfrauenklinik Mannheim, Mannheim
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Caritas - Krankenhaus Saint Josef, Regensburg
  - Klinikum Obergoeltzsch Rodewisch, Rodewisch
  - Klinikum Rosenheim, Rosenheim
  - Klinikum Landkreis Tuttlingen, Tuttlingen
- National Institute of Oncology, Budapest, Hungary
- Tata Memorial Hospital, Mumbai, India
- Italy (12):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Sanitaria di Bolzano, Bolzano
  - Spedali Civili di Brescia, Brescia
  - Ospedale Civile Ramazzini, Carpi
  - European Institute of Oncology, Milan
  - Fondazione Salvatore Maugeri, Pavia
  - Misericordia e Dolce Hospital, Prato
  - Ospedale Civile Rimini, Rimini
  - Istituto Clinico Humanitas, Rozzano
  - Policlinico Universitario Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Waikato Hospital, Hamilton, New Zealand
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Sandton Oncology Centre, Johannesburg, South Africa
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - University Hospital of Linkoping, Linköping
  - Skaraborgs Hospital, Skövde
- Switzerland (13):
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Oncocare Sonnenhof-Klinik Engeriedspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Onkologie-Praxis ZeTup Chur, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale "la Carita", Locarno, Locarno
  - Ospedale Civico, Lugano
  - Ospedale Beata Vergine, Mendrisio
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - UniversitaetsSpital Zuerich, Zurich
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, England
  - Peterborough Hospitals Trust, Peterborough, England
  - South Tyneside District Hospital, South Shields, England

REFERENCES:
- [Background] Francis P, Fleming G, Nasi ML, et al.: Tailored treatment investigations for premenopausal women with endocrine responsive (ER+ and/or PGR+) breast cancer: the SOFT, TEXT, and PERCHE trials. [Abstract] The Breast 12 (Suppl 1): A-P104, S44, 2003.
- [Background] Regan MM, Pagani O, Walley B, Torrisi R, Perez EA, Francis P, Fleming GF, Price KN, Thurlimann B, Maibach R, Castiglione-Gertsch M, Coates AS, Goldhirsch A, Gelber RD; SOFT/TEXT/PERCHE Steering Committee and the International Breast Cancer Study Group. Premenopausal endocrine-responsive early breast cancer: who receives chemotherapy? Ann Oncol. 2008 Jul;19(7):1231-1241. doi: 10.1093/annonc/mdn037. Epub 2008 Mar 5. PMID 18325918
- [Background] Rabaglio M, Ruepp B; Soft/Text/Perche Steering Committee. Death due to liver failure during endocrine therapy for premenopausal breast cancer. Acta Oncol. 2010 Aug;49(6):874-6. doi: 10.3109/0284186X.2010.484813. No abstract available. PMID 20482225
- [Background] Regan MM, Pagani O, Fleming GF, Walley BA, Price KN, Rabaglio M, Maibach R, Ruepp B, Coates AS, Goldhirsch A, Colleoni M, Gelber RD, Francis PA; International Breast Cancer Study; GroupSOFT and TEXT Investigators. Adjuvant treatment of premenopausal women with endocrine-responsive early breast cancer: design of the TEXT and SOFT trials. Breast. 2013 Dec;22(6):1094-100. doi: 10.1016/j.breast.2013.08.009. Epub 2013 Oct 2. PMID 24095609
- [Result] Pagani O, Regan MM, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Perez EA, Ciruelos E, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Pinotti G, Puglisi F, Crivellari D, Ruhstaller T, Winer EP, Rabaglio-Poretti M, Maibach R, Ruepp B, Giobbie-Hurder A, Price KN, Bernhard J, Luo W, Ribi K, Viale G, Coates AS, Gelber RD, Goldhirsch A, Francis PA; TEXT and SOFT Investigators; International Breast Cancer Study Group. Adjuvant exemestane with ovarian suppression in premenopausal breast cancer. N Engl J Med. 2014 Jul 10;371(2):107-18. doi: 10.1056/NEJMoa1404037. Epub 2014 Jun 1. PMID 24881463
- [Result] Pagani O, Walley BA, Fleming GF, Colleoni M, Lang I, Gomez HL, Tondini C, Burstein HJ, Goetz MP, Ciruelos EM, Stearns V, Bonnefoi HR, Martino S, Geyer CE Jr, Chini C, Puglisi F, Spazzapan S, Ruhstaller T, Winer EP, Ruepp B, Loi S, Coates AS, Gelber RD, Goldhirsch A, Regan MM, Francis PA; SOFT and TEXT Investigators and the International Breast Cancer Study Group (a division of ETOP IBCSG Partners Foundation). Adjuvant Exemestane With Ovarian Suppression in Premenopausal Breast Cancer: Long-Term Follow-Up of the Combined TEXT and SOFT Trials. J Clin Oncol. 2023 Mar 1;41(7):1376-1382. doi: 10.1200/JCO.22.01064. Epub 2022 Dec 15. PMID 36521078
- [Derived] O'Regan RM, Ren Y, Zhang Y, Fleming GF, Francis PA, Pagani O, Walley BA, Kammler R, Dell'Orto P, Viale G, Loi S, Colleoni M, Treuner K, Regan MM. Identifying premenopausal patients with early-stage hormone receptor-positive breast cancer at minimal risk of distant recurrence by breast cancer index. Breast. 2026 Jan 29;86:104714. doi: 10.1016/j.breast.2026.104714. Online ahead of print. PMID 41637791
- [Derived] Ribi K, Cole BF, Fleming GF, Walley BA, Francis PA, Abdi E, Burstein HJ, Cheng KL, Chia SKL, Dakhil SR, Davidson NE, Della-Fiorentina SA, Frith AE, Levine E, Lupichuk S, Pritchard K, Salim M, Stearns V, Stewart J, Valero V, van der Westhuizen A, Pagani O, Loi S, Colleoni M, Gelber RD, Goldhirsch A, Coates AS, Regan MM, Bernhard J. Prognostic value of patient-reported depression in women with hormone-responsive early breast cancer in TEXT and SOFT. Cancer. 2025 Oct 1;131(19):e70094. doi: 10.1002/cncr.70094. PMID 40986647
- [Derived] Pagani O, Francis PA, Fleming GF, Walley BA, Viale G, Colleoni M, Lang I, Gomez HL, Tondini C, Pinotti G, Di Leo A, Coates AS, Goldhirsch A, Gelber RD, Regan MM; SOFT and TEXT Investigators and International Breast Cancer Study Group. Absolute Improvements in Freedom From Distant Recurrence to Tailor Adjuvant Endocrine Therapies for Premenopausal Women: Results From TEXT and SOFT. J Clin Oncol. 2020 Apr 20;38(12):1293-1303. doi: 10.1200/JCO.18.01967. Epub 2019 Oct 16. PMID 31618131
- [Derived] Francis PA, Pagani O, Fleming GF, Walley BA, Colleoni M, Lang I, Gomez HL, Tondini C, Ciruelos E, Burstein HJ, Bonnefoi HR, Bellet M, Martino S, Geyer CE Jr, Goetz MP, Stearns V, Pinotti G, Puglisi F, Spazzapan S, Climent MA, Pavesi L, Ruhstaller T, Davidson NE, Coleman R, Debled M, Buchholz S, Ingle JN, Winer EP, Maibach R, Rabaglio-Poretti M, Ruepp B, Di Leo A, Coates AS, Gelber RD, Goldhirsch A, Regan MM; SOFT and TEXT Investigators and the International Breast Cancer Study Group. Tailoring Adjuvant Endocrine Therapy for Premenopausal Breast Cancer. N Engl J Med. 2018 Jul 12;379(2):122-137. doi: 10.1056/NEJMoa1803164. Epub 2018 Jun 4. PMID 29863451
- [Derived] Regan MM, Walley BA, Francis PA, Fleming GF, Lang I, Gomez HL, Colleoni M, Tondini C, Pinotti G, Salim M, Spazzapan S, Parmar V, Ruhstaller T, Abdi EA, Gelber RD, Coates AS, Goldhirsch A, Pagani O. Concurrent and sequential initiation of ovarian function suppression with chemotherapy in premenopausal women with endocrine-responsive early breast cancer: an exploratory analysis of TEXT and SOFT. Ann Oncol. 2017 Sep 1;28(9):2225-2232. doi: 10.1093/annonc/mdx285. PMID 28911092
- [Derived] Johansson H, Gray KP, Pagani O, Regan MM, Viale G, Aristarco V, Macis D, Puccio A, Roux S, Maibach R, Colleoni M, Rabaglio M, Price KN, Coates AS, Gelber RD, Goldhirsch A, Kammler R, Bonanni B, Walley BA; the TEXT principal investigators. Impact of CYP19A1 and ESR1 variants on early-onset side effects during combined endocrine therapy in the TEXT trial. Breast Cancer Res. 2016 Nov 8;18(1):110. doi: 10.1186/s13058-016-0771-8. PMID 27825388
- [Derived] Regan MM, Francis PA, Pagani O, Fleming GF, Walley BA, Viale G, Colleoni M, Lang I, Gomez HL, Tondini C, Pinotti G, Price KN, Coates AS, Goldhirsch A, Gelber RD. Absolute Benefit of Adjuvant Endocrine Therapies for Premenopausal Women With Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer: TEXT and SOFT Trials. J Clin Oncol. 2016 Jul 1;34(19):2221-31. doi: 10.1200/JCO.2015.64.3171. Epub 2016 Apr 4. PMID 27044936
- [Derived] Bernhard J, Luo W, Ribi K, Colleoni M, Burstein HJ, Tondini C, Pinotti G, Spazzapan S, Ruhstaller T, Puglisi F, Pavesi L, Parmar V, Regan MM, Pagani O, Fleming GF, Francis PA, Price KN, Coates AS, Gelber RD, Goldhirsch A, Walley BA. Patient-reported outcomes with adjuvant exemestane versus tamoxifen in premenopausal women with early breast cancer undergoing ovarian suppression (TEXT and SOFT): a combined analysis of two phase 3 randomised trials. Lancet Oncol. 2015 Jul;16(7):848-58. doi: 10.1016/S1470-2045(15)00049-2. Epub 2015 Jun 16. PMID 26092816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2672 patients were randomized between 7Nov03 and 7Apr11 at 182 centers in 15 countries.
Period: Overall Study
Arm/Group | T+OFS | E+OFS
Started | 1334 | 1338
Completed | 1034 | 1026
Not Completed | 300 | 312
Not completed — Adverse Event | 83 | 116
Not completed — Death | 3 | 0
Not completed — Lack of Efficacy | 126 | 78
Not completed — Lost to Follow-up | 45 | 43
Not completed — Withdrawal by Subject | 43 | 75

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population excludes 12 patients who immediately withdrew consent, were at a non-adherent center, or had inadequate documentation of informed consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | T+OFS | E+OFS | Total
Number analyzed (Participants) | 1328 | 1332 | 5320
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  Age: number analyzed (Participants) | 1328 | 1332 | 2660
  Age | 44 [40 to 46] | 43 [39 to 46] | 43 [40 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 1328 | 1332 | 2660
  Female | 1328 | 1332 | 2660
  Male | 0 | 0 | 0
Lymph-node status [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Negative: number analyzed (Participants) | 1328 | 1332 | 2660
    Negative | 52 | 52 | 104
    Positive: number analyzed (Participants) | 1328 | 1332 | 2660
    Positive | 48 | 48 | 96
Tumor size [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    <=2 cm: number analyzed (Participants) | 1328 | 1332 | 2660
    <=2 cm | 60 | 59 | 119
    >=2 cm: number analyzed (Participants) | 1328 | 1332 | 2660
    >=2 cm | 39 | 40 | 79
    unknown: number analyzed (Participants) | 1328 | 1332 | 2660
    unknown | 1 | 1 | 2
Tumor grade [Number; unit: percent of participants] — Tumor grade is the histologic grade according to the BRE method. The method involves assessment of tumor morphology, including tubule formation, nuclear pleomorphism and frequency of mitoses. Grades are recorded according to criteria as 1,2 or 3. Grade 3 is associated with poor prognosis. Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    1: number analyzed (Participants) | 1328 | 1332 | 2660
    1 | 17 | 17 | 34
    2: number analyzed (Participants) | 1328 | 1332 | 2660
    2 | 56 | 55 | 111
    3: number analyzed (Participants) | 1328 | 1332 | 2660
    3 | 26 | 27 | 53
    unknown: number analyzed (Participants) | 1328 | 1332 | 2660
    unknown | 1 | 1 | 2
HER2 status [Number; unit: percent of participants] — Units in this baseline measure reflect the percentage of total participants, rather than number of participants. The total provided does not equal the total number of participants and should not be interpreted as an accurate total of participants.
  percent of participants
    Negative: number analyzed (Participants) | 1328 | 1332 | 2660
    Negative | 87 | 87 | 174
    Positive: number analyzed (Participants) | 1328 | 1332 | 2660
    Positive | 12 | 12 | 24
    Unknown: number analyzed (Participants) | 1328 | 1332 | 2660
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where disease-free survival is defined as the time from randomization to the first appearance of one of the following: invasive breast cancer recurrence at local, regional, or distant site, invasive contralateral breast cancer, second (non-breast) invasive cancer, or death without cancer event; or censored at date of last follow up.
Time Frame: 5-year estimate reported at a median follow-up of 72 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T+OFS | E+OFS
Number analyzed (Participants) | 1328 | 1332
percentage of participants | 87.3 [85.7 to 88.7] | 91.1 [89.7 to 92.3]
Statistical Analysis 1: Comparison: T+OFS vs E+OFS; Test type: Superiority or Other; p = .0002, Log Rank; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.602 to 0.855] — T+OFS is the reference group in the estimation of the hazard ratio

2. Secondary Outcome: Breast Cancer-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where breast cancer-free interval is defined as the time from randomization to the invasive breast cancer recurrence at local, regional, or distant site, or invasive contralateral breast cancer; or censored at date of last follow up.
Time Frame: 5-year estimate reported at a median follow-up of 72 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T+OFS | E+OFS
Number analyzed (Participants) | 1328 | 1332
percentage of participants | 88.8 [87.3 to 90.1] | 92.8 [91.6 to 93.9]
Statistical Analysis 1: Comparison: T+OFS vs E+OFS; Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.664, 95% CI 2-sided [.548 to .804] — T+OFS is the reference group for the estimation of the hazard ratio

3. Secondary Outcome: Distant Recurrence-free Interval
Description: Estimated percentage of patients alive and disease-free at 5 years from randomization, where distant recurrence-free interval is defined as the time from randomization to breast cancer recurrence at a distant site; or censored at date of last follow-up
Time Frame: 5-year estimates reported at a median follow-up of 72 months
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T+OFS | E+OFS
Number analyzed (Participants) | 1328 | 1332
percentage of participants | 92.0 [90.7 to 93.1] | 93.8 [92.7 to 94.8]
Statistical Analysis 1: Comparison: T+OFS vs E+OFS; Test type: Superiority or Other; p = 0.02, Log Rank; Hazard Ratio (HR) = 0.777, 95% CI 2-sided [0.624 to 0.967] — T+OFS was the reference group in the estimation of the hazard ratio

4. Secondary Outcome: Overall Survival
Description: Estimated percentage of patients alive at 8 years from randomization, where overall survival is defined as the time from randomization to death from any cause; or censored at date last known alive.
Time Frame: 8-year estimates, reported at a median follow-up of 9 years
Population: Intention-to-treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T+OFS | E+OFS
Number analyzed (Participants) | 1328 | 1332
percentage of participants | 93.3 [92.1 to 94.3] | 93.4 [92.2 to 94.4]
Statistical Analysis 1: Comparison: T+OFS vs E+OFS; Test type: Superiority; p = 0.84, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.79 to 1.22] — T+OFS was the reference group in the estimation of the hazard ratio

ADVERSE EVENTS:
Time Frame: Assessed every 3 months for the first year, then every 6 months until year 6. Reported at a median follow-up of 72 months.
Description: Targeted adverse events and other grade 3 or higher adverse events were collected on CRFs, regardless of attribution. The safety population EXCLUDES patients who never started protocol-assigned therapy.
Arm/Group | T+OFS | E+OFS
Serious Adverse Events (participants affected / at risk) | 484/1321 | 496/1317
Other Adverse Events (participants affected / at risk) | 1293/1321 | 1298/1317
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T+OFS (N=1321) | E+OFS (N=1317)
Hemolysis (e.g., immune hemolytic anemia, drug related hemolysis, other) (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura or hemolytic uremic syndrome) (Blood and lymphatic system disorders) | 1 | 0
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Hemoglobin (Blood and lymphatic system disorders) | 3 | 2
Cardiac Arrhythmia-Other (Specify) (Cardiac disorders) | 1 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 4
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 3 | 1
Pain - Cardiac/heart (Cardiac disorders) | 0 | 1
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2 | 2
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 2 | 0
Supraventricular and nodal arrhythmia - Supraventricular arrhythmia NOS (Cardiac disorders) | 1 | 0
Supraventricular and nodal arrhythmia - Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Valvular heart disease (Cardiac disorders) | 0 | 1
Auditory/Ear-Other (Specify) (Ear and labyrinth disorders) | 1 | 1
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 2 | 0
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 | 1
Endocrine-Other (Specify) (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 1
Retinopathy (Eye disorders) | 1 | 0
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 | 1
Hemorrhage, GI - Varices (rectal) (Gastrointestinal disorders) | 1 | 0
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 1
Perforation, GI - Duodenum (Gastrointestinal disorders) | 1 | 0
Stricture/stenosis (including anastomotic), GI - Esophagus (Gastrointestinal disorders) | 1 | 0
Ulcer, GI - Stomach (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 0 | 2
Gastrointestinal-Other (Specify) (Gastrointestinal disorders) | 1 | 3
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 9 | 15
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 | 3
Pain - Stomach (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 32 | 41
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 | 0
Death not associated with CTCAE term - Sudden death (General disorders) | 1 | 0
Flu-like syndrome (General disorders) | 1 | 0
Injection site reaction/extravasation changes (General disorders) | 1 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 4
Pain-Other (Specify) (General disorders) | 2 | 0
Obstruction, GI - Gallbladder (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 1
Hepatobiliary/Pancreas-Other (Specify) (Hepatobiliary disorders) | 5 | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 5 | 1
Pain - Gallbladder (Hepatobiliary disorders) | 0 | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 7 | 5
Allergy/Immunology-Other (Specify) (Immune system disorders) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Foreign body (e.g., graft, implant) (Infections and infestations) | 4 | 0
Infection with unknown ANC - Foreign body (e.g., graft, implant, prosthesis, stent) (Infections and infestations) | 1 | 0
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Catheter-related (Infections and infestations) | 0 | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Wound (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Appendix (Infections and infestations) | 1 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Bronchus (Infections and infestations) | 1 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 0 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Joint (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 5 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Middle ear (otitis media) (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Nerve-peripheral (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Pelvis NOS (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Salivary gland (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 8 | 9
Infection with normal ANC or Grade 1 or 2 neutrophils - Small bowel NOS (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Soft tissue NOS (Infections and infestations) | 0 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Stomach (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 0 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Wound (Infections and infestations) | 0 | 2
Infection with unknown ANC - Appendix (Infections and infestations) | 1 | 1
Infection with unknown ANC - Bronchus (Infections and infestations) | 0 | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 2 | 0
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 2 | 4
Infection-Other (Specify) (Infections and infestations) | 4 | 2
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 11 | 18
Intra-operative injury - Ureter (Injury, poisoning and procedural complications) | 0 | 1
Intra-operative injury - Vagina (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 29 | 13
Vessel injury-vein - Extremity-upper (Injury, poisoning and procedural complications) | 0 | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 6 | 3
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 6 | 4
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 0 | 1
Bilirubin (hyperbilirubinemia) (Investigations) | 0 | 1
Carbon monoxide diffusion capacity (DL(co)) (Investigations) | 1 | 0
GGT (gamma-glutamyl transpeptidase) (Investigations) | 2 | 4
INR (International Normalized Ratio of prothrombin time) (Investigations) | 0 | 1
Leukocytes (total WBC) (Investigations) | 0 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 | 2
Weight loss (Investigations) | 1 | 2
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 | 8
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 5 | 8
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-function (Musculoskeletal and connective tissue disorders) | 1 | 1
Lymphedema-related fibrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 | 8
Pain - Back (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 69 | 139
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 | 1
Secondary Malignancy-possibly related to cancer treatment (Specify) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hemorrhage, CNS (Nervous system disorders) | 1 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 9 | 2
Dizziness (Nervous system disorders) | 2 | 3
Memory impairment (Nervous system disorders) | 1 | 1
Neurology-Other (Specify) (Nervous system disorders) | 2 | 4
Neuropathy: cranial - CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 2 | 0
Neuropathy: motor (Nervous system disorders) | 0 | 2
Neuropathy: sensory (Nervous system disorders) | 1 | 0
Pain - Head/headache (Nervous system disorders) | 9 | 11
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 2 | 12
Seizure (Nervous system disorders) | 1 | 1
Syncope (fainting) (Nervous system disorders) | 1 | 4
Vasovagal episode (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 54 | 44
Mood alteration - anxiety (Psychiatric disorders) | 1 | 3
Mood alteration - depression (Psychiatric disorders) | 59 | 51
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 0 | 1
Incontinence, urinary (Renal and urinary disorders) | 3 | 2
Obstruction, GU - Ureter (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Renal/Genitourinary-Other (Specify) (Renal and urinary disorders) | 24 | 7
Hemorrhage, GU - Uterus (Reproductive system and breast disorders) | 0 | 1
Hemorrhage, GU - Vagina (Reproductive system and breast disorders) | 4 | 1
Breast nipple/areolar deformity (Reproductive system and breast disorders) | 0 | 1
Irregular menses (change from baseline) (Reproductive system and breast disorders) | 0 | 1
Pain - Vagina (Reproductive system and breast disorders) | 11 | 33
Sexual/Reproductive Function-Other (Specify) (Reproductive system and breast disorders) | 3 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Obstruction/stenosis of airway - Larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hot flashes/flushes (Vascular disorders) | 149 | 127
Hypertension (Vascular disorders) | 100 | 90
Hypotension (Vascular disorders) | 1 | 0
Vascular-Other (Specify) (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T+OFS (N=1321) | E+OFS (N=1317)
Cardiac-ischemia/infarction (Cardiac disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 446 | 478
Fatigue (asthenia, lethargy, malaise) (General disorders) | 807 | 760
Injection site reaction/extravasation changes (General disorders) | 99 | 86
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 56 | 60
Fracture (Injury, poisoning and procedural complications) | 57 | 82
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 3 | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 30 | 31
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 16 | 17
Osteoporosis (Musculoskeletal and connective tissue disorders) | 388 | 588
Pain - Joint (Musculoskeletal and connective tissue disorders) | 953 | 1030
Hemorrhage, CNS (Nervous system disorders) | 12 | 7
CNS cerebrovascular ischemia (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 738 | 714
Libido (Psychiatric disorders) | 486 | 555
Mood alteration - depression (Psychiatric disorders) | 592 | 610
Incontinence, urinary (Renal and urinary disorders) | 232 | 182
Pain - Vagina (Reproductive system and breast disorders) | 336 | 374
Vaginal dryness (Reproductive system and breast disorders) | 611 | 683
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 752 | 705
Hot flashes/flushes (Vascular disorders) | 1081 | 1076
Hypertension (Vascular disorders) | 179 | 213

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No